CLINICAL TRIAL: NCT00403689
Title: Effects of (1,3), (1,6)-Beta-D-glucan on Insulin Sensitivity and Inflammatory Markers of the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: Danone Research Foundation (Unknown); Leiber Company (Unknown)
Responsible Party: Principal Investigator, Weickert, Martin O., Chief Investigator, German Institute of Human Nutrition
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MOW_bGlucan
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Overweight
Keywords: Increased non-specific inflammatory markers
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- x (Experimental): capsules containing beta glycan
  Interventions: Dietary Supplement: Beta-D-Glucan
- y (Placebo Comparator): capsules containing placebo (waxy maize starch)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Beta-D-Glucan — 1,5 g Beta-D-Glucan daily
  Arms: x
Dietary Supplement: placebo — 1.5 g waxy maize starch daily
  Arms: y

SUMMARY:
Insoluble (1,3),(1,6)-beta-D-glucan from bakers yeast are indigestible polysaccharides. Previous studies indicate that the intake of insoluble dietary fiber is strongly associated with reduced risk of type 2 diabetes and cardiovascular disease. However, the mechanisms leading to this phenomenon are largely unknown.

There are close relations between metabolic and inflammatory pathways, and a number of hormones, cytokines, signal proteins, bioactive lipids, and transcription factors have been shown to be involved in both systems.

Beta-D-glucans have been suggested to play a role as so called biological response modifiers. Studies in animals indicate that even small doses of (1,3),(1,6)-beta-D-glucan may have beneficial effects on immune activity, i.e., by reducing the secretion of inflammatory factors.

The investigators hypothesize that the intake of isolated (1,3), (1,6)-beta-D-glucan from bakers yeast improves inflammatory makers and insulin-sensitivity in overweight subjects with increased C-reactive protein concentrations at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal glucose tolerance (NGT)
* Impaired glucose tolerance (IGT)
* Impaired fasting glucose (IFG)

Exclusion Criteria:

* Any severe cardiac disease
* Liver
* Kidney diseases
* Type 1 or type 2 diabetes
* Chronical and acute inflammatory diseases
* Lipid lowering drugs
* Cortisone
* Antibiotics
* Non-steroidal antiinflammatory drugs
* Including low dose acetylsalicylic acid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Beta-D-glucan induced changes in inflammatory markers, adipokines, and gut hormones. Changes in insulin-sensitivity. | 3 days

SECONDARY OUTCOMES:
Altered gene expression in adipose tissue if changes in primary outcome measures are shown. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin O Weickert, MD, Principal Investigator — German Institute of Human Nutrition; Andreas FH Pfeiffer, Prof, Study Chair — German Institute of Human Nutrition
Locations (1):
- German Institute of Human Nutrition, Department of Clinical Nutrition, Potsdam-Rehbrücke, Nuthetal, Germany

REFERENCES:
- [Result] Kohl A, Gogebakan O, Mohlig M, Osterhoff M, Isken F, Pfeiffer AF, Weickert MO. Increased interleukin-10 but unchanged insulin sensitivity after 4 weeks of (1, 3)(1, 6)-beta-glycan consumption in overweight humans. Nutr Res. 2009 Apr;29(4):248-54. doi: 10.1016/j.nutres.2009.03.002. PMID 19410976
- See also: Related Info — http://www.dife.de